CLINICAL TRIAL: NCT05028621
Title: Exploratory Analysis of the Molecular Basis of Langerhans and Non-Langerhans Cell Histiocytic Neoplasms and Castleman Disease
Brief Title: Molecular Basis of Langerhans and Non-Langerhans Cell Histiocytic Neoplasms and Castleman Disease
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Working on changing study vendor
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE7Z20
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Castleman's Disease (CD); Langerhans Cell Histiocytosis (LCH); Non-Langerhans-Cell Histiocytosis
MeSH Terms: conditions — Castleman Disease; Histiocytosis, Langerhans-Cell; Histiocytosis, Non-Langerhans-Cell | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Genomic analysis (Experimental): When a participant's disorder was diagnosed, blood or tissue specimen was collected. A part of the tissue or blood will be sent to an outside company, Tempus, to be tested for specific genetic changes and the results will be sent back to participants' physician.
  Interventions: Diagnostic Test: Genetic testing

INTERVENTIONS:
Diagnostic Test: Genetic testing — Genetic testing of blood or tissue sample and limited medical information sent to an outside company. Database will link genome sequence data with human trait information, including cancer and other diseases, to be sent to participant's physician.

SUMMARY:
The purpose of this study is to use agnostic genomic evaluation using whole exome sequencing (WES) of a variety of rare hematologic diseases grouped under rare blood diseases and its variants to further elucidate the understanding of the chemistry of these disorders and identify potential actionable mutations that can be targeted with therapies in the context of clinical trials.

DETAILED DESCRIPTION:
The study team will examine genetic changes, also known as mutations, in the DNA of participants' blood, or if applicable, bone marrow specimen. These types of tests are increasingly used by doctors to improve the accuracy of diagnosis and make decisions during care. This study seeks to understand how many patients will benefit from this testing, and in what ways. The results of this portion of the study are placed in the individual's medical record and are communicated back to each participant.

ELIGIBILITY:
Inclusion Criteria:

* Must have histopathologic confirmation of the particular rare hematologic disease.
* Diseases that will be considered as rare hematologic diseases for this study will include the following

  * Langerhans cell histiocytosis (LCH)
  * Erdhiem Chester disease (ECD)
  * Rosai-Dorfman disease (RDD)
  * Miscellaneous histiocytic entities -indeterminate dendritic cell tumor, interdigitating dendritic cell sarcoma, follicular dendritic cell sarcoma, fibroblastic reticular cell tumor
  * Unicentric Castleman disease
  * Multicentric Castleman disease including TAFRO
  * Follicular Dendritic Cell sarcoma (FDCS)
* Newly diagnosed treatment naïve patients as well as patients who received prior therapies (e.g. chemotherapy, targeted therapy, surgery, or radiation) will be included. -Tissue specimens collected within the past 5 yearse will be considered acceptable for study inclusion will include the following
* Collected as part of the evaluation for diagnostic confirmation
* Tissue specimen or extracted DNA (from blood sample) banked in IRB approved tissue repositories and obtained within five years prior to the date of informed consent. -Tissue samples are planned to be collectedfrom previously stored surgical specimens already being stored in pathology lab
* Consent to have germline testing performed in parallel to tumor testingg)Patients willing to receive treatmen

Exclusion Criteria:

* Life expectancy of less than 6months
* Patient unwilling to have germline testing performed on peripheral blood or buccal mucosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of genomic analyses yielding genetic aberrations | Up to 12 months from last participant accrued
  Proportion of genomic analyses yielding actionable genetic aberrations. "Actionable" is defined as a mutation linked to an approved therapy in the particular disease under study or another disease, a known or suspected contraindication to a given therapy, or a clinical trial linked to the alteration

SECONDARY OUTCOMES:
Proportion of genomic analyses yielding actionable genetic aberrations | Up to 12 months from last participant accrued
  Actionable will be defined as a mutation linked to an approved therapy in the particular disease or another disease, a known or suspected contraindication to a given therapy, or a clinical trial linked to the alteration.
Proportion of genomic analyses yielding germline genetic aberrations | Up to 12 months from last participant accrued
Referral rates for genetic counseling for germline mutations | Up to 12 months from last participant accrued
  Number of participants with germline mutations who were referred to genetic counseling through Cancer Genetics for their identified germline mutations
Completion rates of genetic counseling for germline mutations | Up to 12 months from last participant accrued
  Number of participants with germline mutations who were referred to, and underwent (completed) genetic counseling through Cancer Genetics.

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared to maintain patient confidentiality